CLINICAL TRIAL: NCT00199446
Title: A Phase 2, Double-blind, Placebo-controlled, Randomized, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of 40mg/Day KW-6002 (Istradefylline) in Subjects With Restless Legs Syndrome
Brief Title: Study of Istradefylline (KW-6002) for the Treatment of Restless Legs Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-US-201
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Sleep Disorder; Restless Legs Syndrome
Keywords: Sleep -Sleep Disorder; Sleep- Restless Legs Syndrome; Clinical Trial
MeSH Terms: conditions — Sleep Wake Disorders; Restless Legs Syndrome | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
The primary purpose of this study is to evaluate the efficacy, safety, and tolerability of 40 mg per day of istradefylline (KW6002) in patients with Restless Legs Syndrome.

DETAILED DESCRIPTION:
Restless Legs Syndrome (RLS) is a very common neurological disorder with a prevalence of approximately 10% in the adult population. It is characterized by an almost irresistible urge to move the legs, usually accompanied by feelings of intense discomfort. The feelings are usually present while at rest and are temporarily relieved by activity. Symptoms are worse in the evening and at night and lead to profound sleep disturbance and daytime fatigue.

Although a number of therapeutic approaches have been used to treat the symptoms of RLS, none have been universally adopted. While it has been shown that some dopaminergic anti-parkinsonian medications are effective in treating RLS, their use may be somewhat limited by side effects associated with long-term dopaminergic activation. Istradefylline may provide a nondopaminergic approach to the treatment of RLS.

This study will compare the efficacy of 40 mg per day of istradefylline in improving the symptoms of RLS with placebo.

ELIGIBILITY:
Inclusion Criteria:

RLS that is mild to moderate in severity, non-nursing and non-pregnant if female, with an otherwise normal examination.

Exclusion Criteria:

Unable to stop other RLS medication, treatment with excluded medications, abnormal medical status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-07; Primary Completion 2006-08 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in an RLS rating scale score at endpoint (6 weeks of treatment or early discontinuation).

SECONDARY OUTCOMES:
Change from baseline values in an RLS rating scale score, in the a sleepiness scale, in values for Clinical Global Impression, in quality of life, and in actigraphic measurements.
Safety

CONTACTS AND LOCATIONS:
Overall Officials: James Williams, MD, Study Director — Kyowa Kirin, Inc.
Locations (1):
- Kyowa Pharmaceutical Inc., Princeton, New Jersey, United States